CLINICAL TRIAL: NCT01686958
Title: Phase 1 Study: A Prospective, Multi-center, Single Arm Study - Evaluation of the Safety and Feasibility of MRI-guided Transurethral Ultrasound Therapy for the Ablation of Prostate Tissue in Patients With Localized Prostate Cancer
Brief Title: Safety Study of MRI-guided Transurethral Ultrasound Ablation of Prostate Tissue to Treat Localized Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Profound Medical Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOC-10246
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Results first posted 2018-10-25 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; High intensity transurethral ultrasound ablation; MRI-guided; Minimally invasive; Real-time temperature feedback control
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MR-Guided Transurethral US Ablation (Experimental): MR-Guided Transurethral US Ablation of Prostate Tissue
  Interventions: Device: MR-Guided Transurethral US Ablation of Prostate Tissue

INTERVENTIONS:
Device: MR-Guided Transurethral US Ablation of Prostate Tissue — The technology is developed to treat patients with organ confined prostate cancer. The therapeutic endpoint of this technology is thermal coagulation of prostate tissue.
  Other Names: Prostate Ablation Device: PAD-105

SUMMARY:
This study is to evaluate that the magnetic resonance imaging (MRI)-guided transurethral ultrasound therapy system is safe and feasible to ablate prostate tissue in men with localized prostate cancer.

DETAILED DESCRIPTION:
Profound Medical Inc. has developed a novel technology called the MRI-guided transurethral ultrasound therapy system. The technology is developed for patients with organ confined prostate cancer. The therapeutic endpoint of this technology is thermal coagulation of prostate tissue.

The treatment is conducted completely within an MRI suite, which enables real-time temperature images of the heated region to be acquired as the ultrasonic treatment is delivered. Using MRI thermometry during treatment, dynamic temperature feedback control over the intensity of the ultrasound beams and rotation of the Ultrasound Applicator can shape the pattern of thermal coagulation accurately and precisely in the prostate gland, thereby reducing the risk of possible damage to important surrounding anatomy such as the rectum, urinary sphincters, neurovascular bundles and pelvic bone. This coagulation method, therefore, has the potential to have lower complication rates than conventional therapies.

ELIGIBILITY:
Inclusion Criteria:

* Male, age ≥65
* Patient with low-risk, early-stage organ-confined prostate cancer (Stage T1c or T2a, N0, M0).
* Gleason score 6 (3+3)
* Prostate-specific antigen (PSA) ≤ 10 ng/ml
* Eligible for MR imaging (DOC-10252)
* Meets the following criteria on pre-treatment transrectal ultrasound imaging:

  1. No cysts or calcifications > 1.0 cm in size
  2. No evidence of extraprostatic extension or seminal vesicle invasion
  3. Overall prostate size less than 5 cm in sagittal length and less than 7 cm in diameter
* Biopsy confirmed adenocarcinoma of the prostate, performed at least 6 weeks prior to and no more than 6 months prior to the scheduled treatment.
* Eligible for General Anesthesia, as defined in American Society of Anesthesiologists (ASA)
* Normal rectal anatomy and rectal mucosa on digital rectal examination

Exclusion Criteria:

* Bleeding disorder
* Abnormal coagulation and current anticoagulant therapy.
* Acute or chronic Urinary Tract Infection
* Interest in future fertility
* History of allergy relevant medication or other
* History of any other malignancy other than skin cancer
* Patients with peripheral arterial disease with intermittent claudication or Leriches Syndrome
* Prior treatment of the prostate gland
* Prior treatment with 5 alpha reductase inhibitor allowed (not as prostate cancer treatment or prevention) as long as drug has been stopped for minimum 3 months
* History of any major rectal or pelvic surgery
* History of ulcerative colitis or other chronic inflammatory conditions affecting rectum
* History of documented clinical prostatitis requiring therapy within previous 6 months
* History of urethral and bladder outlet disorders, including urethral stricture disease, urethral diverticulae, bladder neck contracture, urethral fistulae which had required prior urethrotomy, urethral stenting, urethroplasty or chronic indwelling urethral catheter
* Patients with artificial urinary sphincter or any penile implant (metallic or non-metallic)
* Neurologic bladder disorders
* Untreated bladder stones
* History of acute urinary retention
* Confirmed or suspected bladder cancer
* Urinary sphincter abnormalities
* Active untreated gross hematuria for any cause
* Post Void Residual (PVR) bladder volume > 250 mL
* Obstructing median lobe enlarged out of proportion to the rest of the prostate and protruding significantly into the bladder

Additional exclusion criteria on file....

Ages: 65 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03-13 (Actual); Primary Completion 2015-03-23 (Actual); Study Completion 2019-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Chin, MD, Principal Investigator — London Health Science Center; James Relle, MD, Principal Investigator — Corewell Health East; Ryan Berglund, MD, Principal Investigator — The Cleveland Clinic; Heinz P Schlemmer, MD, Principal Investigator — German Cancer Research Center
Locations (3):
- William Beaumont Hospital, Royal Oak, Michigan, United States
- London Health Science Centre, London, Ontario, Canada
- German Cancer Research Center (DKFZ), Heidelberg, Germany

REFERENCES:
- [Derived] Chin JL, Billia M, Relle J, Roethke MC, Popeneciu IV, Kuru TH, Hatiboglu G, Mueller-Wolf MB, Motsch J, Romagnoli C, Kassam Z, Harle CC, Hafron J, Nandalur KR, Chronik BA, Burtnyk M, Schlemmer HP, Pahernik S. Magnetic Resonance Imaging-Guided Transurethral Ultrasound Ablation of Prostate Tissue in Patients with Localized Prostate Cancer: A Prospective Phase 1 Clinical Trial. Eur Urol. 2016 Sep;70(3):447-55. doi: 10.1016/j.eururo.2015.12.029. Epub 2016 Jan 6. PMID 26777228

RESULTS

PARTICIPANT FLOW:
Groups:
- MR-Guided Transurethral Ultrasound Ablation of Prostate Tissue: Technology developed to treat patients with organ confined prostate cancer. The therapeutic endpoint of this technology is whole gland ablation.
  Study is a prospective, multi-center, single arm trial conducted in US, Canada and Europe. All subjects received the same treatment.
  Treatment delivery using an investigational medical device, PAD-105, a MRI-guided transurethral ultrasound whole gland prostate ablation.
Period: Overall Study
Arm/Group | MR-Guided Transurethral Ultrasound Ablation of Prostate Tissue
Started | 30
Completed | 29 (No. of patients who completed ALL assessments at 12 months post treatment; 1 pt only had PSA test.)
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Baseline measures were only done for the patients who passed screening and eligibility criteria
Groups:
- MR-Guided Transurethral US Ablation: MR-Guided Transurethral US Ablation of Prostate Tissue
  MR-Guided Transurethral US Ablation of Prostate Tissue: The technology is developed to treat patients with organ confined prostate cancer. The therapeutic endpoint of this technology is thermal coagulation of prescribed prostate tissue.
Arm/Group | MR-Guided Transurethral US Ablation
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Data was collected via a questionnaire completed by the patient at the Baseline Visit. Patients were asked to describe themselves by noting a "X" in one box only. Available options included; White/Caucasian; Black/African-American; Latino/Hispanic' Asian/Pacific Islander; Multi-Racial; Other.
  Participants
    Multi-racial | 1
    White/Caucasian | 29
Region of Enrollment [Number; unit: participants]
  Canada | 12
  United States | 4
  Germany | 14
Subjects with erections sufficient for penetration at Baseline [Count of Participants; unit: Participants] — Erectile dysfunction was defined as a score of 0-1 for Question 2 of the International Index of Erectile Function (IIEF-15). Patients with erections sufficient for penetration had a score greater than or equal to 2.
  Participants | 21

OUTCOME MEASURES:

1. Primary Outcome: Safety - Evaluate the Frequency of Treatment Related Adverse Events
Description: All reported adverse events were recorded. The frequency was measured as the number of study participants who experienced a treatment/device related adverse event after receiving treatment delivery with PAD-105, the investigational device.
Time Frame: 12 months from the Treatment Date
Population: The safety population consists of all subjects who underwent treatment delivery with PAD-105, the investigational medical device.
Measure: Count of Participants; unit: Participants
Groups:
- MR-Guided Transurethral Ultrasound Ablation of Prostate Tissue: The technology is developed to treat patients with organ confined prostate cancer. The therapeutic endpoint of this technology is whole gland ablation.
  Treatment delivery using an investigational medical device, PAD-105, a MRI-guided transurethral ultrasound whole gland prostate ablation.
Arm/Group | MR-Guided Transurethral Ultrasound Ablation of Prostate Tissue
Number analyzed (Participants) | 30
Participants | 30
Statistical Analysis 1: Comparison: MR-Guided Transurethral Ultrasound Ablation of Prostate Tissue; A total of 30 subjects will be accrued to this study and treated with the PAD-105. The sample size is based primarily on feasibility and logistical concerns, however, is sufficiently large to allow the safety objectives to be met. Specifically, with 30 total patients, if no treatment-related grade 4 or 5 adverse events are observed, then a one-sided, 95% confidence interval would have an upper bound of 0.095; Test type: Other — This is a primarily descriptive study, no statistical analysis is planned; however, analyses were performed at the alpha=0.05 level of significance and exact analyses will be used wherever possible; Confidence intervals [CI] will be constructed for outcomes of interest at the alpha=0.05 level of significance, i.e. 95% CI; For continuous outcomes, standard summary statistics will include n, mean, standard deviation, median, minimum and maximum. For categorical data, tables will show n and % of patients

2. Secondary Outcome: Feasibility - Evaluate the Effectiveness of the Investigational System to Thermally Coagulate Prostate Tissue Conforming to the Target Volume With a High Degree of Accuracy and Precision
Description: Conformal thermal coagulation of prostate tissue will be determined quantitatively using measures of targeting accuracy which compare the spatial difference between the target volume and target temperature isotherm determined from MR thermometry images acquired during treatment.
Time Frame: On Treatment Date
Population: The analysis population consists of all subjects who underwent treatment delivery with PAD-105, the investigational medical device.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | MR-Guided Transurethral Ultrasound Ablation of Prostate Tissue
Number analyzed (Participants) | 30
mm
  Thermal ablation accuracy | 0.1 (0.4)
  Thermal ablation precision | 1.3 (0.4)

3. Other Pre Specified Outcome: Treatment Efficacy - Biopsy
Description: Evaluate the effectiveness of the treatment to achieve disease control at 12 months based on biopsy results.
Time Frame: 12 months from the Treatment Date
Population: One patient did not complete the 12-month visit, therefore 29 patients were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | MR-Guided Transurethral Ultrasound Ablation of Prostate Tissue
Number analyzed (Participants) | 29
Participants
  Positive biopsy (clinically significant disease) | 9
  Overall absence of clinically significant disease | 20

4. Other Pre Specified Outcome: Treatment Efficacy - PSA
Description: Based on measurements obtained at each study visit, characterize the pattern of PSA response within the first 12 months following treatment in comparison to baseline.
Time Frame: As per the Study Schedule, measured at 1-month, 3-months, 6-months and 12-months from the Treatment Date compared to Baseline
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | MR-Guided Transurethral Ultrasound Ablation of Prostate Tissue
Number analyzed (Participants) | 30
ng/ml
  PSA @ Baseline | 5.8 [3.8 to 8.0]
  PSA @ 1 month | 0.8 [0.5 to 1.1]
  PSA @ 3 months | 0.9 [0.4 to 1.7]
  PSA @ 6 months | 0.8 [0.4 to 1.1]
  PSA @ 12 months | 0.8 [0.6 to 1.1]

5. Other Pre Specified Outcome: Treatment Efficacy - Quality of Life - Urinary Symptoms
Description: Evaluate quality of life in the first 12 months following Treatment compared to Baseline, using a standardized questionnaire, International Prostate Symptom Score (IPSS), which focuses on urinary symptoms.
  Total Score: 0 - 35 0-7 - mildly symptomatic 8-19 - moderately symptomatic 20-35 - severely symptomatic
Time Frame: Baseline and 12-months post Treatment
Population: One patient did not complete the 12-month visit questionnaire in its entirety, hence overall number of patients analyzed is 29 versus 30 at baseline.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | MR-Guided Transurethral Ultrasound Ablation of Prostate Tissue
Number analyzed (Participants) | 30
units on a scale
  IPSS @ Baseline | 8 [5 to 13]
  IPSS @ 12 months: number analyzed (Participants) | 29
  IPSS @ 12 months | 5 [4 to 7]

6. Other Pre Specified Outcome: Treatment Efficacy - Quality of Life - Erectile Function
Description: Evaluate quality of life in the first 12 months following Treatment compared to Baseline, using a standardized questionnaire, Erectile Function EF domain of the International Index of Erectile Function (IIEF-15), which focuses on erectile symptoms.
  Minimum score value - 0 Maximum score value - 30 A higher score corresponds to a better outcome; lower score indicative of erectile dysfunction
Time Frame: Baseline and 12-months post Treatment
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | MR-Guided Transurethral Ultrasound Ablation of Prostate Tissue
Number analyzed (Participants) | 30
units on a scale
  IIEF-EF-15 @ Baseline | 13 [6 to 28]
  IIEF-EF-15 @ 12 months: number analyzed (Participants) | 29
  IIEF-EF-15 @ 12 months | 13 [5 to 25]

7. Other Pre Specified Outcome: Treatment Efficacy - Quality of Life - Bowel Habits
Description: Evaluate quality of life in the first 12 months following Treatment compared to Baseline, using a standardized questionnaire, Bowel Habits domain of the UCLA Prostate Cancer Index Short Form (UCLA-PCl-SF-BH), which focuses on bowel symptoms.
  Minimum score value - 0 Maximum score value - 100 A higher score corresponds to better outcome
Time Frame: Baseline and 12-months post Treatment
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- MR-Guided Transurethral Ultrasound of Prostate Tissue Ablation: The technology is developed to treat patients with organ confined prostate cancer. The therapeutic endpoint of this technology is whole gland ablation.
  Treatment delivery using an investigational medical device, PAD-105, a MRI-guided transurethral ultrasound whole gland prostate ablation.
Arm/Group | MR-Guided Transurethral Ultrasound of Prostate Tissue Ablation
Number analyzed (Participants) | 30
units on a scale
  UCLA-PCI-SF-BH @ Baseline | 100 [90 to 100]
  UCLA-PCI-SF-BH @ 12 months: number analyzed (Participants) | 29
  UCLA-PCI-SF-BH @ 12 months | 100 [100 to 100]

8. Primary Outcome: Safety - Evaluate the Severity of Treatment Related Adverse Events
Description: Severity of treatment/device related adverse events were evaluated in accordance with the Common Terminology Criteria for Adverse Events (CTCAE) standard (version 4), published by the National Cancer Institute (NCI).
  There was no intraoperative complication, no rectal injury or fistula and no severe urinary incontinence. No Grade 4 (G4) or higher adverse events and only one attributable Grade 3 (G3) event; reported below. The common and significant Grade 1 (G1) and Grade 2 (G2) genitourinary events have also been reported.
Time Frame: 12 months from the Treatment Date
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % of subjects
Arm/Group | MR-Guided Transurethral Ultrasound Ablation of Prostate Tissue
Number analyzed (Participants) | 30
% of subjects
  Hematuria - G1 | 43 [25 to 63]
  Hematuria - G2 | 6.7 [0.8 to 22]
  Urinary tract infection - G2 | 33 [17 to 53]
  Epididymitis - G3 | 3.3 [0.1 to 17]
  Urinary retention - G1 | 10 [2.1 to 27]
  Urinary retention - G2 | 17 [5.6 to 35]
  Obstructive micturition | 10 [2.1 to 27]
  Urinary incontinence - G1 | 3.3 [0.1 to 17]
  Urinary incontinence - G2 | 10 [2.1 to 27]
  Urinary stricture - G1 | 3.3 [0.1 to 17]
  Urinary stricture - G2 | 3.3 [0.1 to 17]

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events were assessed and documented at each follow-up visit. The severity was evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE) standard published by the National Cancer Institute (NCI).
Arm/Group | MR-Guided Transurethral US Ablation
Serious Adverse Events (participants affected / at risk) | 2/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MR-Guided Transurethral US Ablation (N=30)
Epididymitis (Infections and infestations) | 1 — Patient diagnosed with epididymitis on left side, requiring antibiotics. Shortly thereafter patient developed a fever requiring hospital admission with changes to prescribed antibiotics.
Urinary retention (Renal and urinary disorders) | 1 — After removal of suprapubic catheter (SPC) as per protocol, the patient experienced retention and received an urethral catheter, but he continued experiencing retention, hence was hospitalized & required a second SPC.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MR-Guided Transurethral US Ablation (N=30)
Hematuria (Renal and urinary disorders) | 15
Urinary tract infection (Renal and urinary disorders) | 10
Epididymitis (Infections and infestations) | 1
Urinary retention (Renal and urinary disorders) | 8
Urinary incontinence (Renal and urinary disorders) | 4
Urinary stricture (Renal and urinary disorders) | 2
Rectal pain (Gastrointestinal disorders) | 1
Fecal straining (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 3
Bladder inflammation (Renal and urinary disorders) | 1
Bladder irritability (Renal and urinary disorders) | 1
Bladder spasm (Renal and urinary disorders) | 5
Edema: penile and/or scrotal (Renal and urinary disorders) | 5
Edema: testicular (Renal and urinary disorders) | 1
Hemorrhagic cystitis (Renal and urinary disorders) | 1
Increased post void urinary residual in bladder (Renal and urinary disorders) | 2
Nocturia (Renal and urinary disorders) | 2
Obstructive micturition (Renal and urinary disorders) | 3
Penile discharge or bleeding (Renal and urinary disorders) | 10
Prostate anatomical change or discoloration (Renal and urinary disorders) | 7
Prostate inflammation (Renal and urinary disorders) | 1
Prostate tissue sloughing (Renal and urinary disorders) | 1
Scarred urethra (Renal and urinary disorders) | 1
Urethral skin tags (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 10
Urinary hesitancy (Renal and urinary disorders) | 7
Urinary sensation to void (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 12
Urine abnormality (Renal and urinary disorders) | 2
Erectile dysfunction or worsening erectile function (Reproductive system and breast disorders) | 11
Ejaculation disorder (Reproductive system and breast disorders) | 7
Hematospermia (Reproductive system and breast disorders) | 2
Distended abdomen (General disorders) | 1
Ear drainage (General disorders) | 1
Fatigue (General disorders) | 1
Fever (Infections and infestations) | 1
Hematoma or Ecchymosis: Buttock (General disorders) | 1
Hemtoma or Ecchymosis: Femur (General disorders) | 1
Hematoma or Ecchymosis: Sacral bone (General disorders) | 1
Hyperkalemia (General disorders) | 1
Patient movement at onset of treatment (General disorders) | 1
Raised lump: Back (General disorders) | 1
Sore throat (General disorders) | 1
Dysuria (Renal and urinary disorders) | 6
Pain: Back, hips, shoulder, upon catheter removal (General disorders) | 5
Pain: Bladder, penile, perineal, prostate, urethral (Renal and urinary disorders) | 12
Suprapubic Catheter: bleeding around SPC, urine leaking around SPC, blocked SPC, catheter fell out (General disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor will review the publication text within twenty days of receipt, however, Sponsor can request changes if text contains Sponsor's Confidential Information, or text contains information for which the Sponsor wishes to obtain patent protection, whereupon such information will be removed or there will be a delay to the presentation or publication to enable the Sponsor to proceed with patent application for an additional 60 days or until patent application has been filed, whichever is earlier.